CLINICAL TRIAL: NCT00705731
Title: Adherence and the Economics of Colon Cancer Screening
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: A105658; R01CA106773 (NIH); K24DK080941 (NIH); 3R01CA106773-04S1 (NIH)
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Cancer Screening
Keywords: Colorectal cancer (CRC); Colorectal cancer screening; Colonoscopy; Fecal occult blood test (FOBT); Cost-effectiveness
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will compare patient adherence to different colorectal cancer (CRC) screening tests to identify the most cost-effective strategy to decrease mortality from CRC. We hypothesize that different types of tests will have different adherence rates, that these rates will alter the cost-effectiveness analysis, and that we can identify patient variables associated with non-adherence to specific CRC screening strategies.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a significant and preventable disease, yet CRC screening rates remain low. Previous investigators have identified barriers to adherence to CRC screening; however, the majority of data have been retrospectively derived, and the limited data produced from prospective assessment have been limited to fecal occult blood testing (FOBT). Constructs based on the Health Belief Model have been proposed to identify items associated with non-adherence to CRC screening, but prospective validation of this model is lacking. The U.S. Preventive Services Task Force report cites a major cause of uncertainty for calculation of the incremental cost-effectiveness of CRC screening is the deficit in primary data regarding adherence to CRC screening tests, specifically whether heterogeneity exists in screening rates of competing strategies. The Institute of Medicine confirmed the importance of detecting heterogeneity in adherence between strategies, understanding that some strategies currently recommended for CRC screening may be dominated by strategies that achieve greater levels of adherence.

This study aims to determine whether adherence rates to CRC screening are heterogeneous between competing strategies (FOBT and colonoscopy). This study will also prospectively examine domains of the Health Belief Model to identify associations with non-adherence to screening. Adherence rates specific to tested strategies will be incorporated in our existing economic models to compare the incremental cost-effectiveness of competing CRC screening strategies. These data will greatly impact policy decisions regarding resource allocation for CRC screening. It is also expected that future research based on data generated through this project will aim to develop and test interventions that optimize adherence to screening strategies to decrease mortality from CRC.

Procedures:

Patients who are due for CRC screening and meet eligibility requirements are identified through a query of the electronic medical record database at San Francisco General Hospital (SFGH). A research assistant (RA) obtains the PCP's approval to attempt recruitment at the patient's primary care appointment. The PCP discusses CRC screening with the participant during their regularly scheduled appointment.

Availability of CRC screening tests: Because of capacity constraints in the endoscopy unit at SFGH, the screening method for those at average risk of CRC had been limited to annual fecal occult blood testing (FOBT). However, the gastroenterology department initiated a pilot program which allows different primary care clinics to refer average-risk patients for colonoscopy screening in rotating 3-month time-blocks. To ensure the endoscopy unit has sufficient capacity to provide CRC screening via colonoscopy, providers in a given primary care clinic are able to refer their patients for (a) colonoscopy screening, (b) FOBT screening, or (c) a choice of either colonoscopy or FOBT screening, depending on the time block. This is not a study intervention; providers simply recommend that their patients complete a standard CRC screening test, and discuss the option or options available. Patients who decline to participate in the study undergo colorectal cancer screening under the guidance of their primary care provider; the same screening tests are available to those who participate and those who do not.

After giving written informed consent, participants complete an RA-administered 20-minute survey based on constructs of the Health Belief Model. Participants also grant us approval to review their medical records in one year to determine if they complete screening; those without a record of testing are contacted to determine if they completed testing outside of SFGH.

ELIGIBILITY:
Inclusion Criteria:

* Average-risk subjects (no family history of CRC, no personal history of polyps or CRC).
* 50 years of age or greater, but less than 80 years old.
* Due for CRC screening.
* Upcoming appointment scheduled with primary care provider.
* Primary care provider has agreed to refer patients for consideration of enrollment in the study.

Exclusion Criteria:

* Family history of CRC in a first-degree relative.
* Personal history of colonic adenomatous polyps, CRC or inflammatory bowel disease.
* Symptoms for which colonoscopy or sigmoidoscopy would otherwise be performed (hematochezia, new onset diarrhea or constipation, abdominal pain).
* CRC screening current (FOBT within preceding 12 months, flexible sigmoidoscopy or double contrast barium enema within 5 years, or colonoscopy within 10 years).
* Comorbid illness precluding endoscopic evaluation (coronary artery disease with myocardial infarction within 6 months, unstable angina or congestive heart failure, chronic obstructive pulmonary disease requiring home oxygen, other diseases that limit life expectancy to less than 10 years).

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population of users of outpatient primary care clinics at San Francisco General Hospital at average risk for development of colorectal cancer (CRC). Outpatient clinics include the General Medical Clinic, the Family Health Center, and the Positive Health Program (HIV primary care clinic).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Adherence to colorectal cancer (CRC) screening, defined as completion of the screening strategy (the subject agrees to pursue/scheduled by the primary care provider). | one year, and then annually for two more years
  Initial adherence measured at one year following enrollment. We have secured additional study funding that will allow us to extend the follow-up period for two more years, so we will measure programmatic adherence to CRC screening strategy over a 3-year period.

SECONDARY OUTCOMES:
Preventive Intention: Of those who agree to colonoscopy or FOBT, the proportion of patients who have colonoscopy scheduled or take home FOBT cards. | one year
Preventive Behavior: Of the subjects with a positive FOBT result, determine the proportion adhering to the follow-up colonoscopy. | one year
Identification of variables in the survey (based on the Health Belief Model) which are associated with non-adherence to screening. | one yearone year, and then annually for two more years

CONTACTS AND LOCATIONS:
Overall Officials: Hal F Yee, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Inadomi JM, Vijan S, Janz NK, Fagerlin A, Thomas JP, Lin YV, Munoz R, Lau C, Somsouk M, El-Nachef N, Hayward RA. Adherence to colorectal cancer screening: a randomized clinical trial of competing strategies. Arch Intern Med. 2012 Apr 9;172(7):575-82. doi: 10.1001/archinternmed.2012.332. PMID 22493463